CLINICAL TRIAL: NCT06907524
Title: Community-Based Preventative Cardiometabolic Screening and Health Coaching- A Prospective Study
Brief Title: Preventative Screening and Health Coaching in a Food Insecure Population
Acronym: HEALTHCOACH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: The Physicians' Foundation (Unknown)
Responsible Party: Principal Investigator, Daniel Luger, Chairman of Medicine, Rush Oak Park, Cardiovascular Prevention and Clinical Lipidology, Division of Cardiology, Rush University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 24112509; 2024DOH05 (Other Grant/Funding Number: The Physicians' Foundation)
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Cardiovascular Disease Prevention; Cardiometabolic Diseases; Cardiovascular Risk Factor; Cardiovascular Risk Score; Hypertension; Hyperlipidemia; Diabetes; Lifestyle Modification; Health Coaching
Keywords: Cardiovascular Disease Prevention; Cardiometabolic Disease Screening; Hypertension; Hyperlipidemia; Diabetes; Lifestyle Modification; Health Coaching; Cardiovascular Risk Score; Atherosclerotic Cardiovascular Disease Risk Score; Cardiovascular Risk Factor; Cardiometabolic Disease
MeSH Terms: conditions — Hypertension; Hyperlipidemias; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: The described study is a longitudinal study directed at investigating the role of virtual health coaching on mitigation of cardiometabolic disease risk. Patients will be recruited from existing community screening events organized by the Cardiometabolic Health Initiative (CHI). CHI is a mobile screening clinic that provides comprehensive cardiometabolic health screenings to clients of food pantries on the west side of Chicago, Illinois. Eligible patients will be recruited and will receive individualized, virtual health coaching directed at lifestyle modification in order to improve cardiometabolic health.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Patients will receive health coaching sessions, conducted by medical students and overseen by a licensed health coach, directed at individualized lifestyle modification relevant to the patient's cardiometabolic health profile. Patients will receive blood pressure cuffs and will be instructed as to how to measure and keep a log of their blood pressure to be reviewed during health coaching sessions. Sessions will occur biweekly for 1 month followed by the next 2 months. Sessions will last approximately 15 minutes in length. Objective data including blood pressure, point-of-care lipid panel and hemoglobin A1c, 10-year atherosclerotic cardiovascular disease (ASCVD) risk score, as well as surveys regarding depression, sleep apnea, physical activity, social determinants of health, and health literacy will be conducted at the time of study enrollment and at 3 and 6 months of study participation.
  Interventions: Behavioral: Longitudinal, Individualized Health Coaching

INTERVENTIONS:
Behavioral: Longitudinal, Individualized Health Coaching — During in-person events and screening - occurring at the initial screening, 3, and 6 months - patients will receive individualized health coaching by on-site physicians and nurse practitioners specializing in lifestyle medicine. Patients will receive virtual health coaching sessions, conducted by medical students and overseen by a licensed health coach, directed at individualized lifestyle modification relevant to the patient's cardiometabolic health profile. Interventions will include but not limited to: changes in diet, exercise, smoking, and drinking status. Patients will receive blood pressure cuffs and will be instructed as to how to measure and keep a log of their blood pressure to be reviewed during health coaching sessions. Sessions will occur biweekly for the first month and monthly for the following 2 months. Sessions will last approximately 15 minutes in length.

SUMMARY:
The goal of this longitudinal study is to investigate the role of virtual health coaching on mitigation of cardiometabolic disease risk in an underserved, food insecure population. The main questions it aims to answer are:

* Does longitudinal, individualized health coaching directed at lifestyle modification reduce patient 10-year risk of heart attack or stroke?
* Does longitudinal, individualized health coaching directed at lifestyle modification reduce rates of hypertension, hyperlipidemia, and diabetes?
* Does longitudinal, individualized health coaching directed at lifestyle modification improve accessibility to healthcare?

Researchers will investigate the effects of regularly scheduled health coaching sessions on composite cardiometabolic risk profile as well as individual modifiable cardiovascular risk factors.

Participants will:

* Participate in in-person cardiovascular screening, occuring at the time of enrollment, months 3 and 6.
* Engage in virtual health coaching sessions to talk about diet, exercise, weight loss, blood pressure and diabetes control, and accessibility to healthcare
* Keep a log of their blood pressure

DETAILED DESCRIPTION:
ABSTRACT

The high burden of socially driven risk factors prohibits members of low-socioeconomic communities from receiving adequate preventative cardiometabolic care. The Cardiometabolic Health Initiative (CHI) is a health equity organization that deploys mobile, cardiac clinics into local food pantries throughout the West Side of Chicago, engaging a high-risk, food-insecure population. Through physical examinations, point-of-care testing, longitudinal lifestyle counselling and targeted social interventions, CHI brings comprehensive care directly to the disenfranchised. CHI seeks to determine if longitudinal, student-led, health coaching can reduce both measurable cardiometabolic risk factor and social barrier to care. A longitudinal study will assess the effect that structured lifestyle-coaching has on participants' blood lipid levels, hemoglobin A1c, blood pressure, weight, composite 10-year Atherosclerotic Cardiovascular Disease risk score and access to care.

BACKGROUND:

Cardiovascular disease (CVD) remains the leading cause of death in the United States and worldwide.1,2 Social determinants of health (SDoH), including lower socioeconomic status (SES) and race, are associated with a higher prevalence of CVD-related deaths and modifiable CVD risk factors, including hypertension, hyperlipidemia, obesity, smoking and physical inactivity.3-5 Individuals experiencing food insecurity have an elevated risk of CVD compared to individuals who are food secure.7,8 Prior literature has established that lifestyle modifications, such as improved nutrition and increased exercise, along with routine preventative cardiometabolic care, can mitigate CVD risk and related deaths. Despite this, food insecure populations and individuals with lower SES are less likely to receive preventative services due to a myriad of SDOH, such as limited access to providers and financial barriers.5 These disparities underscore the necessity of community-based CVD prevention programs aimed at increasing prevention and detection of modifiable CVD risk factors within high-risk, socially vulnerable populations.

Previous studies have identified the benefit of community-based participatory research (CBPR) in improving cardiometabolic health outcomes. Buchanan et al. conducted regular meetings with tribal councils and home visits over 9 years in 10 Alaskan Native communities and observed significant improvements in CVD risk factors, including blood pressure (BP) and triglyceride levels.9 Interestingly, improvements extended even to community members not included in the study. This effect is thought to be a direct result of CBPR's improvement of overall community health engagement and advocacy.9 Additional studies that partnered with a community advisory board (CAB) also showed improved community health behaviors and outcomes. Notably, a study by Kitzman et al. observed significant weight loss among African American women after utilizing CBPR and a CAB of local pastors.10 In addition to improvements in population health, previous CBPR studies have indicated a positive effect on individual cardiometabolic risk factors. In 2016, Koniak-Griffin et al. observed that amongst a female Latina study population, those who engaged in a culturally tailored Community Health Worker (CHW) led lifestyle behavior intervention showed improved dietary habits, a decrease in waist circumference, and greater awareness of cardiovascular disease risk factors.11 Likewise, Seguin-Fowler et al. developed a 6-month CBPR intervention for rural, medically-underserved women and observed greater improvements in physical activity, healthy diet, and body mass index (BMI) among the intervention group compared to the control group.12 Thus, CBPR incorporates CHWs, community advisors, and community residents to create sustainable community health improvement. Existing literature has proven this model efficacious in improving health within high-risk communities.

However, much of the prior literature on CBPR has focused on testing the effectiveness of group-based lifestyle interventions on lowering the risk for CVD. Only a few studies have analyzed the effect of individualized counseling on mitigating CVD risk. These studies have shown that an individualized approach may be more effective for controlling hypertension. Nakano et al. organized nutritionists to provide intensive nutritional education five times over 12 weeks. This intervention was found to effectively lower BP among hypertensive patients.13 In a study by Ma et al., clinical nurses conducted motivational interviewing eight times over six months and found that antihypertensive medication adherence increased and BP decreased within the intervention group.14 Additionally, no previous research has investigated the efficacy of a CBPR approach in providing individualized counseling to populations experiencing food insecurity, who are at increased risk for CVD.

Research has shown that a CBPR approach in a group setting is effective at mitigating CVD risk, but the literature regarding CBPR within an individualized setting is limited and does not focus on populations experiencing food insecurity in the US.15 Utilizing a CBPR model, the proposed study aims to analyze the impact of individualized, longitudinal lifestyle coaching on mitigating CVD risk amongst food insecure populations in Chicago, Illinois.

OBJECTIVES:

Purpose: The purpose of this study is to investigate the relationship between cardiometabolic health and food insecurity and to analyze the effect of individualized health coaching, directed at lifestyle modification, on cardiometabolic health in an underserved, food insecure population.

Specific Aims:

Specific Aim 1: To determine if preventative screenings and longitudinal health coaching improve the cardiometabolic health of food insecure individuals Specific Aim 2: To analyze the prevalence of cardiometabolic risk factors in food insecure populations in Chicago, Illinois Specific Aim 3: To describe the impact that social determinants of health have on access to care and assess if community-based health screenings can improve accessibility. Specific Aim 4: To develop community-based, preventative health screening protocol that is both culturally sensitive and effective.

Primary Objective:

Evaluate the change in 10-year atherosclerotic cardiovascular disease (ASCVD) risk score after 3 months of longitudinal health coaching.

Secondary Objective:

Analyze change in modifiable cardiovascular risk factors, including blood pressure, blood lipid levels, obesity, physical activity, nutrition, and smoking status following 3 months of longitudinal health coaching.

Determine improvement in barriers to care including access to primary care physicians, social work, or other resources.

Null Hypothesis: Longitudinal health coaching provided to food insecure individuals will have no measurable impact on individuals' composite cardiometabolic risk profile and modifiable cardiovascular risk factors.

RESEARCH METHODS:

Overview of Study Design:

The proposed longitudinal study will assess the effectiveness of health coaching on reducing the risk of cardiometabolic disease. Patients will be recruited from existing community screening events organized by the Cardiometabolic Health Initiative (CHI). CHI is a mobile screening clinic that provides comprehensive cardiometabolic health screenings to clients of food pantries on the West Side of Chicago, Illinois. Eligible patients will receive all services offered at existing, in-person CHI events, including assessment of cardiometabolic risk profile - as determined by measurement of vitals, blood lipids and hemoglobin A1c - in addition to resources offered by community health workers, mental health specialists, and on-site counseling from physicians, nurse practitioners, and health coaches. In addition, patients will receive recurring, virtual, individualized health coaching directed at lifestyle modification. Participants will be reassessed at selected intervals to assess if health coaching and frequent contact with the medical system improved the modifiable cardiovascular risk factors.

Patient Population and Recruitment:

The Cardiometabolic Health Initiative (CHI) is a community service organization with existing strategic partnerships with several food pantries and nonprofit organizations in Chicago. Existing partners include: West Side United, Beyond Hunger, and Harmony Church. At CHI sponsored events, clients of participating food pantries are invited to undergo free, comprehensive cardiometabolic screening. In addition, patients have the opportunity to engage with mental health specialists, community health workers, and health coaching with on-site physicians (including cardiologists and physiatrists), nurse practitioners specializing in lifestyle medicine, and students from Rush University Medical College, College of Nursing, and College of Health Sciences. Individuals will be recruited for participation in the described study from CHI sponsored community screening events.

Vulnerable Populations:

Patients will be recruited at CHI sponsored events conducted at local food pantries in the Chicagoland area. The food pantries serve all individuals, irrespective of social factors, including housing or immigration status. Consequently, the proposed study has the potential to involve several vulnerable populations, such as: undocumented immigrants and refugees, and socioeconomically disadvantaged participants, including the unhoused, uninsured, and low-income. Patients from these populations will not be prevented from participation in the proposed study, nor will their affiliation with any of the aforementioned groups be solicited or documented. The purpose of this study is to analyze an intervention directed towards addressing various barriers to care and all patients who satisfy the inclusion and exclusion criteria will be offered enrollment.

Initial Screening

Following the provision of participant's informed consent, demographic data will be obtained including first and last name, date of birth, sex, race, ethnicity, phone number, zip code. A focused medical history will be obtained, including relevant cardiometabolic comorbidities and medications. Vital signs will be collected: blood pressure, weight, neck and waist circumferences. Blood pressures will be taken in accordance with the American Heart Association (AHA)/American College of Cardiology (ACC) guidelines:

Patients will be seated for 5 minutes with feet firmly on the ground, uncrossed, before the initial measurement. After the initial reading, two additional measurements are taken with one minute in between readings and the blood pressure cuff switched to the opposite arm after each measurement. The last two blood pressure measurements will be averaged as the patient's recorded blood pressure.

Patients will undergo a fingerstick to analyze blood lipid and A1c levels. Point-of-care blood lipid panel will be assessed using the PTS Diagnostics CardioCheck Plus Analyzer and hemoglobin A1c levels will be measured using the Abbott Afinion 2 Analyzer. From this data the patient's 10-year Atherosclerotic Cardiovascular Disease (ASCVD) risk score will be calculated via the MD+Calc ASCVD risk calculator from the AHA/ACC. Additionally, surveys will be completed including the Patient Health Questionnaire 2 (PHQ-2), STOP-BANG, Rapid Assessment of Physical Activity (RAPA), SDOH, and health literacy surveys.

In accordance with existing CHI events, patients will meet with a community health worker (CHW) to discuss any concerns regarding SDOH, including access to a primary care physician (PCP). All patients will have a Rush Epic medical record created, if not already existing, in order for CHWs to document their SDOH screening and any appropriate referrals to social work. For patients without a PCP, a social worker will attempt to contact the patient in order to assist in creating an appointment at a local clinic. Finally, patients will meet with on-site providers, including cardiologists and physiatrists, nurse practitioners specializing in lifestyle medicine, and Rush University students from the Medical College, College of Nursing, and or College of Health Sciences. Providers will discuss participants' screening results and provide appropriate, individualized health coaching. Health coaching will utilize motivational interviewing to provide accessible lifestyle modification recommendations aimed at improving their cardiometabolic health.

Inclusion / Exclusion Criteria:

Inclusion:

Patient is a participant at a CHI sponsored, community screening event Patient provides informed consent and willingness to participate for the duration of the study English or Spanish speaking Age 40-75 years old At least 1 cardiometabolic risk factor at suboptimal level

Defined as one or more of the following at initial screening:

Blood Pressure (BP):

Systolic BP greater than 130mmHg and/or diastolic BP greater than 80mmHg. Obesity: body mass index (BMI) greater than 30 〖kg/m〗^2

Dyslipidemia:

Total cholesterol greater than 200 mg/dL Triglycerides greater than 150 mg/dL Low density lipoprotein (LDL) greater than 130 mg/dL High density lipoprotein (HDL) less than 40 mg/dL in men or less than 50 mg/dL in women Hemoglobin A1c greater than or equal to 5.7% 10-year ASCVD score greater than 5% Access to a telehealth compatible device

Exclusion:

Adults unable to provide informed consent or unwilling to participate for study duration Speaks language other than English or Spanish Younger than 40 years old or older than 75 years old All cardiometabolic risk factors at optimal levels No telehealth compatible device Pregnant patients

Consent Process:

If the patient satisfies all eligibility criteria, written consent for participation in the study will be obtained. Of note, patient participation at CHI sponsored events requires patient signed written consent detailing a patient's willingness to have their vitals and a blood sample collected for the purposes of cardiometabolic screening and counseling. Written consent forms detailing the study protocol, purpose, and patient participation, written in English or Spanish as appropriate, will be given to the patient and explained in detail. Following provision of informed consent, patients will be eligible to participate in study sanctioned screening and health coaching. Patients will be able to withdraw consent at any time, resulting in the patient removal from the study.

STUDY PROTOCOL:

Following initial screening and enrollment, patients will be instructed on how to participate in virtual health coaching utilizing telehealth. Initially, patients will receive individual health coaching sessions biweekly for the first month.

Sessions will be conducted by Rush University students who have completed a specific training program in motivational interviewing led by a licensed health coach. Sessions will last approximately 15 minutes in length. Attempts will be made to standardize the health coaching process through drafted protocols directed at cardiometabolic risk factors. Nonetheless, individualized coaching and planning will be specific and unique to each patient's lifestyle and social considerations. As part of the health coaching, each patient will receive a blood pressure cuff. Patients will be instructed how to accurately measure their blood pressure and keep a log to be reviewed at coaching sessions. After the first month, the interval of health coaching sessions will be extended to monthly for an additional 2 months.

As previously described, patients will participate in the initial screening prior to enrollment in the study. Data collected at the time of screening will include: first and last name, date of birth, sex, race, ethnicity, phone number, zip code, focused medical history including relevant cardiometabolic comorbidities and medications, blood pressure, weight, neck and waist circumferences, point-of-care lipid panel and hemoglobin A1c, 10-year ASCVD risk score, PHQ-2, STOP-BANG, RAPA, SDOH, and health literacy surveys. Following enrollment, patients' cardiometabolic risk profile will be reassessed at 3 and 6 months of study participation at which time the aforementioned data will be recollected to assess for changes in cardiometabolic health.

SAMPLE SIZE:

Power analysis for this study was deferred. At this time, prevalence of cardiometabolic risk factors in a food insecure population are not well reported in the literature. Due to the finite pool of patients who participate in CHI community screening events and satisfy the inclusion and exclusion criteria, all eligible patients will be screened and offered the opportunity to enroll with the understanding that the study may be insufficiently powered. Based on attendance of previous CHI monthly events, we expect to enroll a total of 200 patients.

ELIGIBILITY:
Inclusion:

Patient is a participant at a CHI sponsored, community screening event Patient provides informed consent and willingness to participate for the duration of the study English or Spanish speaking Age 40-75 years old At least 1 cardiometabolic risk factor at suboptimal level

Defined as one or more of the following at initial screening:

Blood Pressure (BP):

Systolic BP greater than 130mmHg and/or diastolic BP greater than 80mmHg. Obesity: body mass index (BMI) greater than 30 〖kg/m〗^2

Dyslipidemia:

Total cholesterol greater than 200 mg/dL Triglycerides greater than 150 mg/dL Low density lipoprotein (LDL) greater than 130 mg/dL High density lipoprotein (HDL) less than 40 mg/dL in men or less than 50 mg/dL in women Hemoglobin A1c greater than or equal to 5.7% 10-year ASCVD score greater than 5% Access to a telehealth compatible device

Exclusion:

Adults unable to provide informed consent or unwilling to participate for study duration Speaks language other than English or Spanish Younger than 40 years old or older than 75 years old All cardiometabolic risk factors at optimal levels No telehealth compatible device Pregnant patients

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
10 - Year Atherosclerotic Cardiovascular Disease Risk Score | From enrollment to the end of study participation at 6 months.
  Study data collected during in-person screening - occuring at the initial screening, 3 and 6 month rescreening - will be utilized to calculate the patient's 10-year Atherosclerotic Cardiovascular Disease (ASCVD) risk via the MD+ Calc ASCVD risk calculator from the American Heart Association (AHA)/American College of Cardiology (ACC).

SECONDARY OUTCOMES:
Depression - Patient Health Questionnaire - 2 (PHQ2) | From enrollment to the end of study participation at 6 months.
  During each in-person screening - initial screening, 3, and 6 month rescreening - patients will be screened for depression using the Patient Health Questionnaire - 2 (PHQ2). Patients who screen positive for depressive symptoms will be referred to on-site mental health specialists for additional resources and care.
Sleep Apnea - STOP-BANG | From enrollment to the end of study participation at 6 months.
  Patients will be screened for sleep apnea at each in-person event - including the initial screening, 3, and 6 month rescreening - using the STOP-BANG survey.
Point-of-care Hemoglobin A1c | From enrollment to the end of study participation at 6 months.
  Patients will undergo a fingerstick to analyze hemoglobin A1c levels using the Abbott Afinion 2 Analyzer. A1c will be measured at the initial screening, 3, and 6 month rescreening.
Point-of-care Blood Lipid Level | From enrollment to the end of study participation at 6 months.
  Patients will undergo a fingerstick to measure a point-of-care blood lipid panel using the PTS Diagnostics CardioCheck Plus Analyzer. Measured data will include: total cholesterol, triglycerides, low-density lipoprotein (LDL), and high-density lipoprotein (HDL). Lipid levels will be measured at the initial screening, 3, and 6 month rescreening.
Blood Pressure | From enrollment to the end of study participation at 6 months.
  Blood pressure will be assessed in accordance with the American Heart Association (AHA)/American College of Cardiology (ACC) guidelines: Patients will be seated for 5 minutes with feet firmly on the ground, uncrossed, before the initial measurement. After the initial reading, two additional measurements are taken with one minute in between readings and the blood pressure cuff switched to the opposite arm after each measurement. The last two blood pressure measurements will be averaged as the patient's recorded blood pressure. Blood pressure will be assessed at the initial screening, 3, and 6 month rescreening. Additionally, patients will be provided blood pressure cuffs and will be directed during health coaching sessions to measure their blood pressure and complete a log to track their measurements.
Physical Activity Level - The Rapid Assessment of Physical Activity (RAPA) Survey | From enrollment to the end of study participation at 6 months.
  Patients will be screened for physical activity levels at each in-person event - including the initial screening, 3, and 6 month rescreening - using The Rapid Assessment of Physical Activity (RAPA) survey.
Accessibility to Healthcare | From enrollment to the end of study participation at 6 months.
  At each in-person event - initial screening, 3, and 6 month rescreening - patients will have the opportunity to meet with licensed community health workers (CHW). CHWs will assess patients' accessibility to healthcare and provide referrals to social workers to help facilitate patients obtaining a primary care physician (PCP). Accessibility to healthcare will be measured by the proportion of patients who have a PCP prior to study intervention as compared to following the completion of participation in the study.
Assessment of Social Determinants of Health | From enrollment to the end of study participation at 6 months.
  Study participants will be screened at each in-person event - initial screening, 3, and 6 month rescreening - for social determinants of health (SDOH). SDOH surveys will be administered by licensed community health workers and will assess for difficulties with finances, transportation, housing, access to food, healthcare, and insurance, physical and emotional safety. Participant's response to SDOH surveys prior to study intervention, throughout the study, and following completion of participation in the study will be assessed.
Assessment of Health Literacy | From enrollment to the end of study participation at 6 months.
  During each in-person study activity - including initial screening, 3, and 6 month rescreening - patients will be presented with a health literacy survey. The survey will assess the patient's diet and knowledge of basic health conditions associated with cardiometabolic health. Patients' responses to the survey prior to intervention, during the study, and following completion of participation in the study will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Luger, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Appel LJ, Champagne CM, Harsha DW, Cooper LS, Obarzanek E, Elmer PJ, Stevens VJ, Vollmer WM, Lin PH, Svetkey LP, Stedman SW, Young DR; Writing Group of the PREMIER Collaborative Research Group. Effects of comprehensive lifestyle modification on blood pressure control: main results of the PREMIER clinical trial. JAMA. 2003 Apr 23-30;289(16):2083-93. doi: 10.1001/jama.289.16.2083. PMID 12709466
- [Background] Soltani D, Azizi B, Behnoush AH, Meysamie A, Aein A, Nayebirad S, Vasheghani-Farahani A, Akbari Sari A. Is lifestyle modification with individual face-to-face education and counseling more effective than usual care for controlling hypertension? A systematic review and meta-analysis of randomized controlled trials. Health Educ Res. 2023 Sep 20;38(5):490-512. doi: 10.1093/her/cyad028. PMID 37450326
- [Background] Ma C, Zhou Y, Zhou W, Huang C. Evaluation of the effect of motivational interviewing counselling on hypertension care. Patient Educ Couns. 2014 May;95(2):231-7. doi: 10.1016/j.pec.2014.01.011. Epub 2014 Jan 30. PMID 24530144
- [Background] Nakano M, Eguchi K, Sato T, Onoguchi A, Hoshide S, Kario K. Effect of Intensive Salt-Restriction Education on Clinic, Home, and Ambulatory Blood Pressure Levels in Treated Hypertensive Patients During a 3-Month Education Period. J Clin Hypertens (Greenwich). 2016 May;18(5):385-92. doi: 10.1111/jch.12770. Epub 2016 Jan 6. PMID 26732187
- [Background] Seguin-Fowler RA, Strogatz D, Graham ML, Eldridge GD, Marshall GA, Folta SC, Pullyblank K, Nelson ME, Paul L. The Strong Hearts, Healthy Communities Program 2.0: An RCT Examining Effects on Simple 7. Am J Prev Med. 2020 Jul;59(1):32-40. doi: 10.1016/j.amepre.2020.01.027. Epub 2020 May 7. PMID 32389532
- [Background] Koniak-Griffin D, Brecht ML, Takayanagi S, Villegas J, Melendrez M, Balcazar H. A community health worker-led lifestyle behavior intervention for Latina (Hispanic) women: feasibility and outcomes of a randomized controlled trial. Int J Nurs Stud. 2015 Jan;52(1):75-87. doi: 10.1016/j.ijnurstu.2014.09.005. Epub 2014 Sep 22. PMID 25307195
- [Background] Kitzman H, Mamun A, Dodgen L, Slater D, King G, King A, Slater JL, DeHaven M. Better Me Within Randomized Trial: Faith-Based Diabetes Prevention Program for Weight Loss in African American Women. Am J Health Promot. 2021 Feb;35(2):202-213. doi: 10.1177/0890117120958545. Epub 2020 Sep 18. PMID 32945175
- [Background] Buchanan Z, Hopkins SE, Ryman TK, Austin MA, Wiener HW, Tiwari HK, Klejka JA, Boyer BB, Fohner AE. Electronic health record reveals community-level cardiometabolic health benefits associated with 10 years of community-based participatory research. Public Health. 2024 Jul;232:38-44. doi: 10.1016/j.puhe.2024.04.010. Epub 2024 May 10. PMID 38733959
- [Background] Liu Y, Eicher-Miller HA. Food Insecurity and Cardiovascular Disease Risk. Curr Atheroscler Rep. 2021 Mar 27;23(6):24. doi: 10.1007/s11883-021-00923-6. PMID 33772668
- [Background] Kris-Etherton PM, Petersen KS, Velarde G, Barnard ND, Miller M, Ros E, O'Keefe JH, Williams K Sr, Horn LV, Na M, Shay C, Douglass P, Katz DL, Freeman AM. Barriers, Opportunities, and Challenges in Addressing Disparities in Diet-Related Cardiovascular Disease in the United States. J Am Heart Assoc. 2020 Apr 7;9(7):e014433. doi: 10.1161/JAHA.119.014433. Epub 2020 Mar 23. PMID 32200727
- [Background] Powell-Wiley TM, Baumer Y, Baah FO, Baez AS, Farmer N, Mahlobo CT, Pita MA, Potharaju KA, Tamura K, Wallen GR. Social Determinants of Cardiovascular Disease. Circ Res. 2022 Mar 4;130(5):782-799. doi: 10.1161/CIRCRESAHA.121.319811. Epub 2022 Mar 3. PMID 35239404
- [Background] Shahu A, Okunrintemi V, Tibuakuu M, Khan SU, Gulati M, Marvel F, Blumenthal RS, Michos ED. Income disparity and utilization of cardiovascular preventive care services among U.S. adults. Am J Prev Cardiol. 2021 Nov 6;8:100286. doi: 10.1016/j.ajpc.2021.100286. eCollection 2021 Dec. PMID 34816144
- [Background] Kim YJ, Kim S, An J, Volgman AS, Nazir NT. Impact of the COVID-19 pandemic on cardiovascular disease mortality in a major metropolitan area. Am Heart J Plus. 2022 Jun;18:100173. doi: 10.1016/j.ahjo.2022.100173. Epub 2022 Jul 13. PMID 35856067
- [Background] Woodruff RC, Tong X, Khan SS, Shah NS, Jackson SL, Loustalot F, Vaughan AS. Trends in Cardiovascular Disease Mortality Rates and Excess Deaths, 2010-2022. Am J Prev Med. 2024 Apr;66(4):582-589. doi: 10.1016/j.amepre.2023.11.009. Epub 2023 Nov 14. PMID 37972797
- [Background] Ahmad FB, Anderson RN. The Leading Causes of Death in the US for 2020. JAMA. 2021 May 11;325(18):1829-1830. doi: 10.1001/jama.2021.5469. No abstract available. PMID 33787821